CLINICAL TRIAL: NCT04040478
Title: Transcutaneous Monitoring of Oxygen and Carbon Dioxide in Surgical Patients for the Detection of Peripheral Tissue Hypoxia and Hypercapnia
Brief Title: Transcutaneous Monitoring of Oxygen and Carbon Dioxide in Surgical Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Radiometer Medical ApS (Industry)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, Head of research, Principal investigator, ass. professor, Rigshospitalet, Denmark
Other Study IDs: TCM study
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Transcutaneous Monitoring; Microcirculation; Peripheral Perfusion; Tissue Metabolism
MeSH Terms: interventions — Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abdominal: 80 patients undergoing surgery for abdominal cancer. Data review for interim analysis will be conducted after the participation of 40 patients to evaluate the requirement for further enrollment.
  Interventions: Device: Transcutaneous monitoring
- Vascular: 20 patients undergoing femoral endarterectomy.
  Interventions: Device: Transcutaneous monitoring

INTERVENTIONS:
Device: Transcutaneous monitoring — Transcutaneous monitoring of oxygen and carbon dioxide by using Radiometer TCM5 flex monitor with 3 electrodes on the patient.
  Abdominal patients are monitored for 4 hours during surgery and for 2 hours in the Post-Anesthesia Care Unit. Arterial blood gasses are drawn from the arterial line 4 times during surgery and 4 times after surgery.
  Patients undergoing vascular surgery are monitored for up to 4 hours during surgery.

SUMMARY:
The study will investigate if non-invasive continuous transcutaneous blood gas monitoring can detect tissue perfusion and hypoxemia and the relation to other circulatory parameters such as pulse, blood pressure, cardiac output and arterial saturation.

DETAILED DESCRIPTION:
Macro circulatory parameters such as cardiac output, mean arterial pressure and arterial oxygen saturation are used to monitor the hemodynamic function and tissue perfusion in surgical patients. Though none of the methods are directly monitoring changes in the metabolism of the tissue. Arterial blood gas analysis is used as the golden standard for the detection of metabolic disturbances before, during and after surgery. Disadvantages of the method are 1) the fact that the technique is invasive to the patient, 2) that the method measures the "total gas" (each tissue's contribution to the blood gas in the total circulating blood) and 3) that the methods only provide a snapshot of the patient's blood gas status. Transcutaneous monitoring can be used as a continuous monitoring of the underlying tissue's carbon dioxide and oxygen levels in patients. The method is already used in neonates as a surrogate for the arterial blood gas analysis. Reduced tissue oxygenation due to inadequate perfusion, will initiate an anaerobic tissue metabolism resulting in low oxygen levels and high carbon dioxide levels. The transcutaneous monitoring can therefore potentially be used to detect tissue hypoxia and become a direct measurement of the underlying tissue metabolism.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery for abdominal cancer
* patients undergoing femoral endarterectomy

Exclusion Criteria:

* patients not able to give a informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to Rigshospitalet due to surgery for abdominal cancer (Whipple procedure) and vascular surgery (femoral endarterectomy)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Changes in tcpO2 and tcpCO2 compared to changes in cardiac output, perfusion index and arterial paO2 and paCO2 | 6 hours
  Percentage changes in tcpO2 and tcpCO2 compared to percentage changes in cardiac output, perfusion index and arterial blood gas analysis of paO2 and paCO2
Changes in tcpO2 and tcpCO2 before, during and after the arterial clamping during the surgery. | 6 hours
  Changes in tcpO2 and tcpCO2 before arterial clamping vs after arterial clamping in the leg undergoing surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eske Aasvang, MD phD DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Sigvardt E, Rasmussen SM, Eiberg JP, Sorensen HBD, Meyhoff CS, Aasvang EK. Transcutaneous blood gas monitoring and tissue perfusion during common femoral thromboendarterectomy. Scand J Clin Lab Invest. 2022 Jul;82(4):334-340. doi: 10.1080/00365513.2022.2092900. Epub 2022 Jun 29. PMID 35767233